CLINICAL TRIAL: NCT05310942
Title: Comparing the Non Invasive Cardiometry With Ultrasound Guided Inferior Vena Cava Collapsibility for Evaluation of Fluid Responsiveness in Septic Patient; Randomized Clinical Trials
Brief Title: Non Invasive Evaluation of Fluid Responsiveness in Septic Patient
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ebtehal Shaheen, assisstant lecturer at faculty of medicine, Benha University
Other Study IDs: MD17-12-2021
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Septic Shock
Keywords: fluid responsiveness; cardiometry; IVC collapsibility
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: The fluid management of patients in this group will be assessed by IVC collapsibility index (IVC CI) calculated by ultrasound through maximum IVC diameter - minimum IVC diameter divided by maximum diameter then multiplied by 100. If it is less than 50% means that the patient is volume non- depleted while if it is more than 50% means the reverse.
- B: All patients in this group with sepsis will be evaluated by the electrical cardiometry monitor.

SUMMARY:
The study aims to evaluate the accuracy of fluid responsiveness assessment with non-invasive cardiometry compared to ultrasound guided inferior vena cava (IVC) collapsibility for management of critically ill septic patients with hemodynamic instability.

DETAILED DESCRIPTION:
Prospective Randomized observational comparative single blinded study will be conducted at intensive care unit at Benha University Hospitals after obtaining approval of the ethical committee and informed written consent from first degree relatives will be issued. The blindness will be performed to the patients.

The study will be conducted according to CONSORT 2010 statement. Enrolment of eligible patients will occur within 8 h of meeting the criteria for septic shock. All patients will be randomized using the computer-generated software of randomization and sealed closed envelopes to allocate them to one of two groups (30 patients each). Routine measurements and investigations will be taken at admission to intensive care unit; history, vital signs, routine laboratory investigation.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I and II
2. Age 18-65 years old of both genders.
3. Fulfilment criteria of sepsis as defined according to the standard Surviving Sepsis Campaign criteria using the Sequential (sepsis-related) Organ Failure Assessment (SOFA) score (SOFA score ≥ 2 indicated organ dysfunction).
4. Patients within 8 h of meeting the criteria for septic shock.

Exclusion Criteria:

1. Lack of consent
2. Age below 18 and above 65 years old.
3. acute coronary syndrome
4. major cardiac dysrhythmia,
5. valvular or congenital heart disease
6. Massive bilateral pleural effusion
7. Severe anaemia
8. End-stage kidney disease (ESKD) patients with Creatinine clearance (CrCl) <50ml/min.
9. Child B and Child C hepatic patients
10. impaired systolic function according to the ejection fraction (EF) (EF < 40% indicated impaired systolic function)
11. Severe ARDS (acute respiratory distress syndrome).
12. Tense ascites
13. Mechanical ventilation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolment of eligible patients will occur within 8 h of meeting the criteria for septic shock. All patients will be randomized using the computer-generated software of randomization and sealed closed envelopes to allocate them to one of two groups (30 patients each). Routine measurements and investigations will be taken at admission to intensive care unit; history, vital signs, routine laboratory investigation.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness | 2 years
  The study primary outcome will be the cardiac index determined by the non-invasive cardiometry in correlation with ultrasound guided IVC collapsibility index to determine which is more effective in prediction of fluid responsiveness.

SECONDARY OUTCOMES:
total infused fluid from ICU arrival till the goal is achieved | 2 years
total dose of vasopressor and inotrope taken during ICU stay period | 2 years
time to weaning of vasopressors and inotropes | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No